CLINICAL TRIAL: NCT02503514
Title: Autoimmune Paradoxical Reactions in IBD Longitudinal Cohort - APRIL Cohort
Brief Title: Autoimmune Paradoxical Reactions in IBD Longitudinal Cohort
Acronym: APRIL
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0167
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Inflammatory Bowel Diseases; Crohns Disease; Ulcerative Colitis; Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Subjects will have blood drawn (10 mL EDTA tube, 10mL Serum Separator, and a 6 mL EDTA tube)at their baseline visit. If a subject experiences a paradoxical reaction they will a repeat of the blood draw done at their baseline visit.
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: Inflammatory bowel disease patients undergoing treatment with varying biologic agents will be evaluated for incidences of paradoxical immune reactions, the risk factors associated with those paradoxical immune reactions, and whether the paradoxical immune reactions and their associated risk factors differ based on formulation of biologic agent.

Participants: All adults (≥18 year) with confirmed IBD on a biologic agent or with plans to initiate treatment in 1 month

Procedures (methods): Subjects undergoing treatment with a biologic agent will be followed indefinitely for paradoxical immune reactions. Data will be collected at baseline as well as serum and plasma for banking. Subjects will be followed at 6 month intervals either via email, telephone interviews or at the time of clinic follow-up visits. In the event of a de-novo paradoxical reaction, specific information will be collected from sites in an event capture form, with data abstracted from routine clinical care for the paradoxical reaction. Subjects will continue to be followed every 3 months after the event via email, telephone contact to determine whether resolution and/or recurrence occurred, and to determine any changes in medical therapy. Serum and plasma will be re-collected at the time of first event for comparison to baseline samples and to samples from controls (those on biologics without study documented paradoxical immune reactions). At resolution of the event, patient will return to 6 month follow up schedule. Subjects can discontinue and/or fail a particular biologic treatment; therefore they will also be followed for paradoxical immune reactions, on any new biologic treatment they undergo while in the study.

DETAILED DESCRIPTION:
Inclusion/Exclusion Criteria: All adults (≥18 year) with confirmed IBD on a biologic agent or with plans to initiate this within 1 month (defined as any anti-TNF, natalizumab, vedolizumab or ustekinumab) will be enrolled into a prospective cohort (initially in a pilot setting at 5 sites, later with full funding involving all sites of the CRA). Individuals with current biologic use will be included (i.e. prevalent users), with records collected as to time of initial biologic start, and prior specific formulations. Ideally, new initiators of biologic agents will be recruited at the visit where the decision is made to start a biologic agent. Those with a prior history of one of the 4 described paradoxical outcomes associated with a biologic agent will also be included as prevalent cases in order to increase the sample size, with appropriate clinical information collected per medical record. All data on prevalent cases will be entered historically prospective follow up with still occur to ensure that paradoxical reaction does not recur.

Exposures: Data will be collected at baseline including demographic and disease specific factors, concomitant medications, laboratory data, as well as serum and plasma for banking.

Follow up: Individuals will be followed at 6 month intervals either via email, telephone interviews or at the time of clinic follow-up visits. Data event forms for outcomes occurring at any point during follow up will be collected real-time in clinic, or if triggered by standard follow-up at 6 months.

Outcome of paradoxical immune reaction: Outcomes are defined as a) psoriaform skin lesion, b) drug-induced lupus c) demyelinating disorder or d) vasculitis. In the event of a de-novo paradoxical reaction, specific information will be collected from sites in an event capture form, with data abstracted from routine clinical care for the paradoxical reaction. Medical records will be obtained confirming the response, with copies of pathology (dermatologic biopsy)or radiology (MRI) reports when applicable. For specific event capture forms. Individuals will continue to be followed every 3 months after the outcome via telephone contact to determine whether resolution and/or recurrence occurred and changes in medical therapy. At resolution of the event, patient will return to 6 month follow up. Serum and plasma will also be re-collected at the time of first outcome in cases for exposure to baseline samples and to those of controls (those on biologics without paradoxical immune reaction). Serum and plasma will be collected at the time of event diagnosis, when possible (within 2 months). If not possible, blood draw can be "missed" in circumstances where patient is not seen in clinic in this window.

Timeline for study contacts:

The top timeline is for an individual who does not develop an event, baseline in-person consent and serum collection, contact every 6 months for telephone contact visit or follow up visit during the time of routine clinic follow-up. The bottom line is for someone who does develop an event, with closer follow-up until event resolution, and repeat serum collection. Contacts therefore range from 3-6 months, with the vast majority having follow up at 6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign informed consent.
* Adults (male or female) with confirmed IBD diagnosed by routine clinical, radiographic, endoscopic and pathological criteria.
* Adults age 18 or older.
* Adults on a new biologic agent or with plans to initiate a biologic agent, within 1 month for the treatment of their IBD.

Exclusion Criteria:

* Inability to understand and sign informed consent.
* Inability to confirm diagnosis of IBD from medical records
* Inability to confirm time of initial biologic start, and prior specific formulations from medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with confirmed IBD on a biologic agent or with plans to initiate this within 1 month.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with specific paradoxical Adverse Events Using Biologic therapies as a part of routine care for the treatment of IBD | 1 year
  Investigator will assess autoimmune reactions such as skin lesions (psoriasis), vasculitis, demyelinating disorders or drug-induced lupus in patients on biologic therapies for IBD. These reactions have been described as "paradoxical inflammation."

CONTACTS AND LOCATIONS:
Overall Officials: Millie D Long, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill- CGIBD, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Benchimol EI, Cook SF, Erichsen R, Long MD, Bernstein CN, Wong J, Carroll CF, Froslev T, Sampson T, Kappelman MD. International variation in medication prescription rates among elderly patients with inflammatory bowel disease. J Crohns Colitis. 2013 Dec;7(11):878-89. doi: 10.1016/j.crohns.2012.09.001. Epub 2012 Sep 25. PMID 23018106
- [Background] van Deen WK, van Oijen MG, Myers KD, Centeno A, Howard W, Choi JM, Roth BE, McLaughlin EM, Hollander D, Wong-Swanson B, Sack J, Ong MK, Ha CY, Esrailian E, Hommes DW. A nationwide 2010-2012 analysis of U.S. health care utilization in inflammatory bowel diseases. Inflamm Bowel Dis. 2014 Oct;20(10):1747-53. doi: 10.1097/MIB.0000000000000139. PMID 25137415
- [Background] Cleynen I, Vermeire S. Paradoxical inflammation induced by anti-TNF agents in patients with IBD. Nat Rev Gastroenterol Hepatol. 2012 Sep;9(9):496-503. doi: 10.1038/nrgastro.2012.125. Epub 2012 Jul 3. PMID 22751454
- [Background] Fiorino G, Danese S, Pariente B, Allez M. Paradoxical immune-mediated inflammation in inflammatory bowel disease patients receiving anti-TNF-alpha agents. Autoimmun Rev. 2014 Jan;13(1):15-9. doi: 10.1016/j.autrev.2013.06.005. Epub 2013 Jun 15. PMID 23777821
- [Background] Rahier JF, Buche S, Peyrin-Biroulet L, Bouhnik Y, Duclos B, Louis E, Papay P, Allez M, Cosnes J, Cortot A, Laharie D, Reimund JM, Lemann M, Delaporte E, Colombel JF; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif (GETAID). Severe skin lesions cause patients with inflammatory bowel disease to discontinue anti-tumor necrosis factor therapy. Clin Gastroenterol Hepatol. 2010 Dec;8(12):1048-55. doi: 10.1016/j.cgh.2010.07.022. Epub 2010 Aug 20. PMID 20728573
- [Background] Afzali A, Wheat CL, Hu JK, Olerud JE, Lee SD. The association of psoriasiform rash with anti-tumor necrosis factor (anti-TNF) therapy in inflammatory bowel disease: a single academic center case series. J Crohns Colitis. 2014 Jun;8(6):480-8. doi: 10.1016/j.crohns.2013.10.013. Epub 2013 Nov 21. PMID 24268978
- [Background] Baumgart DC, Grittner U, Steingraber A, Azzaro M, Philipp S. Frequency, phenotype, outcome, and therapeutic impact of skin reactions following initiation of adalimumab therapy: experience from a consecutive cohort of inflammatory bowel disease patients. Inflamm Bowel Dis. 2011 Dec;17(12):2512-20. doi: 10.1002/ibd.21643. Epub 2011 Feb 23. PMID 21351201
- [Background] Cullen G, Kroshinsky D, Cheifetz AS, Korzenik JR. Psoriasis associated with anti-tumour necrosis factor therapy in inflammatory bowel disease: a new series and a review of 120 cases from the literature. Aliment Pharmacol Ther. 2011 Dec;34(11-12):1318-27. doi: 10.1111/j.1365-2036.2011.04866.x. Epub 2011 Sep 29. PMID 21957906
- [Background] Denadai R, Teixeira FV, Steinwurz F, Romiti R, Saad-Hossne R. Induction or exacerbation of psoriatic lesions during anti-TNF-alpha therapy for inflammatory bowel disease: a systematic literature review based on 222 cases. J Crohns Colitis. 2013 Aug;7(7):517-24. doi: 10.1016/j.crohns.2012.08.007. Epub 2012 Sep 7. PMID 22960136
- [Background] Guerra I, Algaba A, Perez-Calle JL, Chaparro M, Marin-Jimenez I, Garcia-Castellanos R, Gonzalez-Lama Y, Lopez-Sanroman A, Mancenido N, Martinez-Montiel P, Quintanilla E, Taxonera C, Villafruela M, Romero-Mate A, Lopez-Serrano P, Gisbert JP, Bermejo F. Induction of psoriasis with anti-TNF agents in patients with inflammatory bowel disease: a report of 21 cases. J Crohns Colitis. 2012 Jun;6(5):518-23. doi: 10.1016/j.crohns.2011.10.007. Epub 2011 Nov 13. PMID 22398059
- [Background] Sherlock ME, Walters T, Tabbers MM, Frost K, Zachos M, Muise A, Pope E, Griffiths AM. Infliximab-induced psoriasis and psoriasiform skin lesions in pediatric Crohn disease and a potential association with IL-23 receptor polymorphisms. J Pediatr Gastroenterol Nutr. 2013 May;56(5):512-8. doi: 10.1097/MPG.0b013e31828390ba. PMID 23274341
- [Background] Buisson A, Cuny JF, Barbaud A, Schmutz JL, Bigard MA, Gueant JL, Peyrin-Biroulet L. Methotrexate for psoriasiform lesions associated with anti-tumour necrosis factor therapy in inflammatory bowel disease. Aliment Pharmacol Ther. 2012 May;35(10):1175-80. doi: 10.1111/j.1365-2036.2012.05082.x. Epub 2012 Apr 2. PMID 22469155
- [Background] Torres J, Buche S, Delaporte E, Colombel JF. Skin side effects of inflammatory bowel disease therapy. Inflamm Bowel Dis. 2013 Apr;19(5):1086-98. doi: 10.1097/MIB.0b013e3182802c07. PMID 23474780
- [Background] Niess JH, Danese S. Anti-TNF and skin inflammation in IBD: a new paradox in gastroenterology? Gut. 2014 Apr;63(4):533-5. doi: 10.1136/gutjnl-2013-304683. Epub 2013 Apr 9. No abstract available. PMID 23570743
- [Background] Moran GW, Lim AW, Bailey JL, Dubeau MF, Leung Y, Devlin SM, Novak K, Kaplan GG, Iacucci M, Seow C, Martin L, Panaccione R, Ghosh S. Review article: dermatological complications of immunosuppressive and anti-TNF therapy in inflammatory bowel disease. Aliment Pharmacol Ther. 2013 Nov;38(9):1002-24. doi: 10.1111/apt.12491. Epub 2013 Sep 25. PMID 24099467
- [Background] Tillack C, Ehmann LM, Friedrich M, Laubender RP, Papay P, Vogelsang H, Stallhofer J, Beigel F, Bedynek A, Wetzke M, Maier H, Koburger M, Wagner J, Glas J, Diegelmann J, Koglin S, Dombrowski Y, Schauber J, Wollenberg A, Brand S. Anti-TNF antibody-induced psoriasiform skin lesions in patients with inflammatory bowel disease are characterised by interferon-gamma-expressing Th1 cells and IL-17A/IL-22-expressing Th17 cells and respond to anti-IL-12/IL-23 antibody treatment. Gut. 2014 Apr;63(4):567-77. doi: 10.1136/gutjnl-2012-302853. Epub 2013 Mar 6. PMID 23468464
- [Background] Perez-Alvarez R, Perez-de-Lis M, Ramos-Casals M; BIOGEAS study group. Biologics-induced autoimmune diseases. Curr Opin Rheumatol. 2013 Jan;25(1):56-64. doi: 10.1097/BOR.0b013e32835b1366. PMID 23114587
- [Background] Soto Lopes MS, Trope BM, Rochedo Rodriguez MP, Grynszpan RL, Cuzzi T, Ramos-E-Silva M. Paradoxical Reaction to Golimumab: Tumor Necrosis Factor alpha Inhibitor Inducing Psoriasis Pustulosa. Case Rep Dermatol. 2013 Nov 7;5(3):326-31. doi: 10.1159/000350930. eCollection 2013. PMID 24348382
- [Background] Harrison MJ, Dixon WG, Watson KD, King Y, Groves R, Hyrich KL, Symmons DP; British Society for Rheumatology Biologics Register Control Centre Consortium; BSRBR. Rates of new-onset psoriasis in patients with rheumatoid arthritis receiving anti-tumour necrosis factor alpha therapy: results from the British Society for Rheumatology Biologics Register. Ann Rheum Dis. 2009 Feb;68(2):209-15. doi: 10.1136/ard.2007.087288. Epub 2008 Apr 2. PMID 18385277
- [Background] Schmitt J, Rosumeck S, Thomaschewski G, Sporbeck B, Haufe E, Nast A. Efficacy and safety of systemic treatments for moderate-to-severe psoriasis: meta-analysis of randomized controlled trials. Br J Dermatol. 2014 Feb;170(2):274-303. doi: 10.1111/bjd.12663. PMID 24131260
- [Background] Schiff MH, Burmester GR, Kent JD, Pangan AL, Kupper H, Fitzpatrick SB, Donovan C. Safety analyses of adalimumab (HUMIRA) in global clinical trials and US postmarketing surveillance of patients with rheumatoid arthritis. Ann Rheum Dis. 2006 Jul;65(7):889-94. doi: 10.1136/ard.2005.043166. Epub 2006 Jan 26. PMID 16439435
- [Background] Ramos-Casals M, Roberto-Perez-Alvarez, Diaz-Lagares C, Cuadrado MJ, Khamashta MA; BIOGEAS Study Group. Autoimmune diseases induced by biological agents: a double-edged sword? Autoimmun Rev. 2010 Jan;9(3):188-93. doi: 10.1016/j.autrev.2009.10.003. Epub 2009 Oct 23. PMID 19854301
- [Background] Yanai H, Shuster D, Calabrese E, Mlynarsky L, Tumuluri S, Cohen RD. The incidence and predictors of lupus-like reaction in patients with IBD treated with anti-TNF therapies. Inflamm Bowel Dis. 2013 Dec;19(13):2778-86. doi: 10.1097/01.MIB.0000435435.91988.b6. PMID 24185311
- [Background] Singh S, Kumar N, Loftus EV Jr, Kane SV. Neurologic complications in patients with inflammatory bowel disease: increasing relevance in the era of biologics. Inflamm Bowel Dis. 2013 Mar-Apr;19(4):864-72. doi: 10.1002/ibd.23011. PMID 22552994
- [Background] Stubgen JP. Tumor necrosis factor-alpha antagonists and neuropathy. Muscle Nerve. 2008 Mar;37(3):281-92. doi: 10.1002/mus.20924. PMID 18041052
- [Background] Mohan N, Edwards ET, Cupps TR, Oliverio PJ, Sandberg G, Crayton H, Richert JR, Siegel JN. Demyelination occurring during anti-tumor necrosis factor alpha therapy for inflammatory arthritides. Arthritis Rheum. 2001 Dec;44(12):2862-9. doi: 10.1002/1529-0131(200112)44:123.0.co;2-w. PMID 11762947
- [Background] Mohan N, Edwards ET, Cupps TR, Slifman N, Lee JH, Siegel JN, Braun MM. Leukocytoclastic vasculitis associated with tumor necrosis factor-alpha blocking agents. J Rheumatol. 2004 Oct;31(10):1955-8. PMID 15468359